CLINICAL TRIAL: NCT04632303
Title: Early Palliative Care for Patients With Advanced Pancreatic Cancer (EarlyCarePan).
Brief Title: Early Palliative Care for Patients With Advanced Pancreatic Cancer.
Acronym: EarlyCarePan
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inna Chen, MD (Other)
Collaborators: Bispebjerg Hospital (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other); Vejle Hospital (Other); Zealand University Hospital (Other); Hillerod Hospital, Denmark (Other); Herning Hospital (Other)
Responsible Party: Sponsor-Investigator, Inna Chen, MD, Senior physician, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GI 2031
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Early palliative care; Specialized palliative care
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Palliative Care (Experimental): Baseline palliative care visit within 10 calendar days of registration/randomization and palliative care visits (either at clinic or at home) or phone calls (if a visit is not feasible) at least every four weeks throughout the patient's life. Referral to exercise training and nutritional specialist.
  Interventions: Other: Early Palliative Care
- Standard Care Arm (No Intervention): Palliative care visit only upon request from attending oncologist(s) or patient/family.

INTERVENTIONS:
Other: Early Palliative Care — Baseline palliative care visit Palliative care visits/calls at least every 4 weeks throughout life and additionally upon request Referral to exercise training Referral to nutritional specialist
  Arms: Early Palliative Care

SUMMARY:
Pancreatic adenocarcinoma is one of the deadliest cancers. Patients with pancreatic cancer experience marked physical suffering, psychological distress and resource-demanding care at the end-of-life. Therefore, an urgent need exists to evaluate the early specialized palliative care model in a comparative study and across multiple care settings to define quality of life and survival benefits in patients with pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma is one of the deadliest cancers. Approximately half of the patients diagnosed with advanced pancreatic cancer die within 2 months from the diagnosis. Patients eligible for systemic treatment have a median survival of less than one year and often receive limited benefit from chemotherapy, usually with progression of disease after only a few months of treatment. Patients with pancreatic cancer experience marked physical suffering, psychological distress and resource-demanding care at the end-of-life. Complications such as pain, fatigue, malnutrition, cachexia, exocrine insufficiency and diagnosis itself lead to a poor quality of life and are associated with high rates of depression and anxiety.

These invalidating symptoms are best alleviated by attachment to specialized palliative care and by starting this support early in the course of the disease and not just in the terminal phase. Early implementation of specialized palliative care is not a standard of care in Denmark.

Thus, an urgent need exists to evaluate the early, integrated palliative care model in a comparative study and across multiple care settings to define quality of life and survival benefits for patients with pancreatic cancer in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females (aged 18 and over)
* Confirmed by cytology or histology incurable PDAC who are planned to receive medical care for cancer in the first-line setting at the enrolling institution within ≤ 2 weeks
* Written informed consent before any study procedures
* Performance status: ECOG 0-2
* Ability to read and respond to questions or able to complete questions with minimal assistance required from an interpreter or family member
* Planning to receive all medical care for cancer at the enrolling institution.

Exclusion Criteria:

* Patients who are already receiving care from the palliative care service are not eligible for participation in the study
* Exhibiting signs of overt psychopathology or cognitive dysfunction
* Any medical condition that the Investigator considers significant to compromise the safety of the patient or that impairs the interpretation of study assessments
* Patient participating in another interventional study during the surveillance period. This is only relevant for studies that might interfere with the intervention. Participation in protocols related only to treatment will not preclude participation in the present study. Cases of doubt will be settled by the protocol responsible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Adjusted mean change in global health status/QoL score at 12 weeks | 12 weeks
  Adjusted mean change from baseline in global health status/QoL score from the EORTC QLQ-C30 questionnaire at 12 weeks.

SECONDARY OUTCOMES:
Overall survival | 1 year
  Overall survival after randomization, defined as the time from randomization to death from any cause.
Adjusted mean change from baseline in global health status/QoL at 6 and 24 weeks. | 24 weeks
  Adjusted mean change from baseline in global health status/QoL score from the EORTC QLQ-C30 questionnaire at 6 and 24 weeks.
Adjusted mean change from baseline in functional and symptom scales at 6, 12 and 24 weeks | 24 weeks
  Adjusted mean change from baseline in functional and symptom scales from the EORTC QLQ-C30 questionnaire at 6, 12 and 24 weeks.
Chemotherapy dose intensity. | 24 weeks
  Chemotherapy dose intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Nissen, MD, Principal Investigator — Herlev & Gentofte Hospital
Locations (1):
- Herlev & Gentofte University Hospital, Denmark, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No